CLINICAL TRIAL: NCT01142505
Title: Parent-determined Oral Montelukast Therapy for Preschool Wheeze With Stratification for Arachidonate-5-Lipoxygenase (ALOX5) Promoter Genotype
Brief Title: Wheeze and Intermittent Treatment
Acronym: WAIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: University of Aberdeen (Other); University of Leicester (Other)
Responsible Party: Principal Investigator, Jonathan Grigg, Professor of Paediatric Respiratory Medicine, Queen Mary University of London
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08/43/03; 2009-015626-11 (EudraCT Number)
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Wheezing
Keywords: wheeze; preschool; leukotriene; montelukast; 5-lipoxygenase
MeSH Terms: conditions — Respiratory Sounds | interventions — Mannitol; montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients in the placebo arm will be given an inactive version of the investigational medical product formed of the excipient mannitol (which is coated with the active drug montelukast in the active comparator arm)
  Interventions: Drug: Mannitol
- Montelukast (Active Comparator): Patients in the active arm will be given an active version of the investigational medical product formed of the inactive excipient mannitol with a coating of active drug montelukast.
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Mannitol — 4mg once daily granules for 10 days, given orally alone or with cold or warm food from the onset of a cold or wheezing attack.
  Other Names: Pearlitol SD 200
  Arms: Placebo
Drug: Montelukast — 4mg once daily granules for 10 days, given orally alone or with cold or warm food from the onset of a cold or wheezing attack
  Other Names: Singulair
  Arms: Montelukast

SUMMARY:
The clinical aim of this trial is to assess whether intermittent montelukast is an effective treatment strategy in preschool wheeze. The mechanisms aim of the trial is to determine whether there is a genetically highly-responsive subgroup of children. In designing this trial the investigators have incorporated several novel aspects. First, parents will be able to adjust the use of oral montelukast to their child's symptoms. This allows the investigators to recruit both "episodic" and "multi trigger" patterns of preschool wheeze - and control for any change in wheeze pattern during the trial. Second, before the investigators issue the trial medication, the investigators will assess children's leukotriene genes, focusing primarily on a gene called ALOX5. This ALOX5 "stratification" step will ensure that an equal number of potentially "treatment-responsive" children receive the active drug (montelukast) and the dummy medicine - and the equal numbers will help the investigators to assess the role of ALOX5. For the trial, the investigators will first recruit 1,300 children with a history of preschool wheeze, then divide them into the group with "responsive" and "less responsive" genes by their ALOX5 status. The investigators will then issue parents with the trial medication; 50% will be given montelukast and 50% will be given dummy medication. Parents will start the trial medication whenever their child develops a cold, and stop the medication when wheeze resolve. Parents will also be able to give the trial medication for wheeze between colds. Over the 12 month trial period, the investigators will assess the number of unscheduled attendances to a medical practitioner for wheeze for each child. At the end of the trial, the investigators will determine whether montelukast is effective then whether there is a difference in response to montelukast between the 2 ALOX5 gene groups.

At the same time, the investigators will measure many other genes that may influence response to montelukast, as well as the amount of leukotrienes that are excreted in the urine before and during attacks. Using these results, the investigators will be able to both inform national treatment policy, and develop new concepts on the mechanism of preschool wheeze that will inform the development of new therapies. Since children will continue to receive "normal" inhaled therapy, there are no ethical issues in giving a dummy medicine to half of the 1300 children to be recruited. The study will be the largest trial in wheezy preschool children to date, and may open up genetic testing in preschool wheeze.

DETAILED DESCRIPTION:
Background

A quarter of all UK children will have at least one attack of wheeze during the preschool period (1 to 5 years of age). Severe attacks of wheeze in these young children are usually triggered by viral-colds. The majority of affected children will only wheeze with colds, although these attacks may be severe and repeated resulting in GP attendances and hospital admissions. This pattern of wheeze is called "episodic" preschool wheeze. A minority of preschool children wheeze both with and between colds - a pattern that is called "multi-trigger" preschool wheeze. In real life this distinction is blurred, with preschool children changing their pattern of wheeze over time. What is clear is that asthma therapies that are effective in older children with classical "allergic" asthma may not necessarily be effective in preschool wheeze. For example, although a short-course of oral steroids is very effective in treating attacks of wheeze in school age children with "allergic" asthma, the investigators have shown in 2 major trials that a short course of oral steroids does not reduce the severity of attacks of preschool wheeze.

Recently, montelukast, an oral medicine that blocks a substance (leukotriene) that narrows the breathing tubes, has shown promise in preschool wheeze. However, to date, only modest benefits have been reported when large groups of children have been studied. One explanation for this, is that a significant proportion of preschool children do not respond to montelukast, but there is a subgroup who are genetically programmed to respond very well. Recent analysis of trials of montelukast suggests that this responsive subgroup may be defined by variations in leukotriene-producing genes. Thus an understanding of the role of leukotriene genes and leukotriene production in preschool wheeze may better target montelukast treatment in this age group, and inform the development of new therapies.

Trial Description

The clinical aim of this trial is to assess whether intermittent montelukast is an effective treatment strategy in preschool wheeze. The mechanisms aim of the trial is to determine whether there is a genetically highly-responsive subgroup of children. In designing this trial the investigators have incorporated several novel aspects. First, parents will be able to adjust the use of oral montelukast to their child's symptoms. This allows us to recruit both "episodic" and "multi trigger" patterns of preschool wheeze - and control for any change in wheeze pattern during the trial. Second, before the investigators issue the trial medication, the investigators will assess children's leukotriene genes, focusing primarily on a gene called ALOX5. This ALOX5 "stratification" step will ensure that an equal number of potentially "treatment-responsive" children receive the active drug (montelukast) and the dummy medicine - and the equal numbers will help us to assess the role of ALOX5. For the trial, the investigators will first recruit 1,300 children with a history of preschool wheeze, then divide them into the group with "responsive" and "less responsive" genes by their ALOX5 status. The investigators will then issue parents with the trial medication; 50% will be given montelukast and 50% will be given dummy medication. Parents will start the trial medication whenever their child develops a cold, and stop the medication when wheeze resolve. Parents will also be able to give the trial medication for wheeze between colds. Over the 12 month trial period, the investigators will assess the number of unscheduled attendances to a medical practitioner for wheeze for each child. At the end of the trial, the investigators will determine whether montelukast is effective then whether there is a difference in response to montelukast between the 2 ALOX5 gene groups.

At the same time, the investigators will measure many other genes that may influence response to montelukast, as well as the amount of leukotrienes that are excreted in the urine before and during attacks. Using these results, the investigators will be able to both inform national treatment policy, and develop new concepts on the mechanism of preschool wheeze that will inform the development of new therapies. Since children will continue to receive "normal" inhaled therapy, there are no ethical issues in giving a dummy medicine to half of the 1300 children to be recruited. The study will be the largest trial in wheezy preschool children to date, and may open up genetic testing in preschool wheeze.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 10 months and ≤ 5 years old on the day of the first dose of Investigational Medicinal Product
* two or more attacks of parent-reported wheeze
* at least one attack with wheeze validated by a clinician
* the most recent attack within the last 3 months
* contactable by telephone and able to attend one face-to-face review for issue of Investigational Medicinal Product
* parent or guardian able to give written informed consent for their child to participate in the study

Exclusion Criteria:

* any other chronic respiratory condition diagnosed by a clinician including structural airway abnormality (e.g. floppy larynx) and cystic fibrosis
* any chronic condition that increases vulnerability to respiratory tract infection such as severe developmental delay with feeding difficulty
* history of neonatal chronic lung disease
* current continuous oral montelukast therapy
* in a trial using an Investigational Medicinal Product in the previous 3 months prior to recruitment

Ages: 10 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1358 (Actual)
Dates: Start 2010-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Need for unscheduled medical attention | 12 months
  Number of times a child attends for an unscheduled medical opinion with respiratory problems over a 12 month period, as confirmed from medical records.

SECONDARY OUTCOMES:
Number of admissions to hospital | 12 months
Duration of admissions to hospital | 12 months
Number of unscheduled GP consultations for wheeze | 12 months
  The number of times a child is brought to his primary care/family doctor with wheeze
Duration of wheezy episodes | 12 months
  The duration of wheezy episodes as recorded by parents on their diary cards.
Severity of episodes by diary card | 12 months
  The severity of wheeze episodes as recorded in parent diary cards
Parent's overall impression of efficacy of Investigational Medicinal Product | 12 months
  Parent's overall impression of efficacy of Investigational Medicinal Product as recorded in diary cards.
Time to first attack of wheeze | 12 months
  Time to first attack of wheeze as recorded in parent diary card and researcher phonecalls.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Grigg, BSc MBBS MD, Principal Investigator — Queen Mary University of London
Locations (1):
- Barts and the London NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Grigg J, Whitehouse A, Pandya H, Turner S, Griffiths CJ, Vulliamy T, T Walton R, Price DB, Sanak M, Holloway JW, Noimark L, Lesosky M, Brugha R, Koh L, Nwokoro C. Urinary prostanoids in preschool wheeze. Eur Respir J. 2017 Feb 2;49(2):1601390. doi: 10.1183/13993003.01390-2016. Print 2017 Feb. No abstract available. PMID 28153869
- [Derived] Nwokoro C, Pandya H, Turner S, Eldridge S, Griffiths CJ, Vulliamy T, Price D, Sanak M, Holloway JW, Brugha R, Koh L, Dickson I, Rutterford C, Grigg J. Intermittent montelukast in children aged 10 months to 5 years with wheeze (WAIT trial): a multicentre, randomised, placebo-controlled trial. Lancet Respir Med. 2014 Oct;2(10):796-803. doi: 10.1016/S2213-2600(14)70186-9. Epub 2014 Sep 8. PMID 25212745